CLINICAL TRIAL: NCT06659523
Title: Exploring Unconventional Plant-Derived Metabolites for Glycemic Control: the Case of Pomegranate
Acronym: EXPLORER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regina Menezes (Other)
Collaborators: Universidade LusÃ³fona de Humanidades e Tecnologias (Unknown)
Responsible Party: Sponsor-Investigator, Regina Menezes, Principal Investigator, Lusofona University
Organization: Lusofona University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CE.ECTS/P05-24
Record Dates: First submitted 2024-08-07; First posted 2024-10-26 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Prediabetes
Keywords: prediabetes; Food supplement; beta-cell function; IAPP; Urolithins
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Supplement Intervention Group (Experimental): 31 healthy individuals, male and female, were recruted at one family health unit, and randomly assigned to the intervention group, and were given for 12 weeks of one daily dose of 1.5 g powdered capsules of EPS.
  Interventions: Dietary Supplement: EPS supplement intervention
- Placebo Group (Placebo Comparator): 29 individuals with pre-diabetes, male and female, were recruted at one family health unit, and randomly assigned to the intervention group, and were given for 12 weeks of one daily dose of placebo supplement (cellulose).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: EPS supplement intervention — 31 healthy individuals, male and female, were recruted at one family health unit, and randomly assigned to the intervention group, and were given for 12 weeks of one daily dose of 1.5 g powdered capsules of EPS.
  Arms: Supplement Intervention Group
Dietary Supplement: Placebo — 29 healthy individuals, male and female, were recruted at one family health unit, and randomly assigned to the placebo group, and were given for 12 weeks of one daily dose of placebo.
  Arms: Placebo Group

SUMMARY:
The EXPLORER study will investigate whether supplementation with a pomegranate extract rich in ellagitannins is able to improve well-being and metabolic health in individuals without diabetes. The aim is to establish for the first time an association between the intake of ellagitanninsa and glycaemic control, the processing/aggregation of IAPP (a protein associated with diabetes), the state of the intestinal microbiota and circulating levels of urolithin B (a small bioavailable molecule resulting from the metabolism of ellagitannins).

This is a 12-week pilot study that is double-blind (neither participants nor researchers know who gets the treatment) and placebo-controlled (some people will receive a non-active substance). It will involve volunteers who do not have diabetes.

Phase 1 - Recruitment: Volunteers without diabetes, who are patients at a family health unit, will be recruited. Participants will provide informed consent and information such as sociodemographic and biochemical data.

Phase 2 - Intervention: The recruited individuals will be divided into two groups: one receiving the pomegranate extract supplement (intervention group) and the other receiving a placebo. In total, 60 participants will take part in the study.

DETAILED DESCRIPTION:
A double-blinded, randomized, placebo-controlled pilot study was designed to assess the effect of Ellagitannins Pomegranate Supplements (EPS) in metabolic health of participants.

Participants will be recruited at the family health unit USF São Martinho de Alcabideche from the grouping of health centres ACES Cascais, and the study will be conducted according to universal bioethical principles.

At least 60 individuals with pre-diabetes will be included in the study. After the fulfilment of the inclusion criteria, they will be randomly assigned to the intervention group (IG) and the placebo group (PG). Equal distribution of gender, age and BMI will be ensured between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Individuals without diabetes
* Both sexes
* Aged between 18 and 65
* Body Mass Index (BMI) less than 29.9 kg/m2
* Fasting plasma glucose levels below 126 mg/dL
* Haemoglobin A1C levels between 5.7 - 6.5%

Exclusion Criteria:

* Not agreeing to take part in the study
* BMI>30 kg/m2
* Being diagnosed with diabetes
* Having any type of cognitive disorder
* Using anti-diabetic medication
* Alcohol or drug abuse
* Pomegranate allergy
* Regular use of food supplements
* Difficulty swallowing tablets
* Being on, or planning to be on during the study period, a different diet than usual
* Pregnancy, planning to become pregnant during the study, breastfeeding 1 year before or during the study
* Oncological, cardiac, hepatic, renal, thyroid or other endocrine diseases
* Medical or social conditions that may affect adherence
* Participating in another study at the same time.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Targeted metabolites - urolithins profiling | 12 weeks
  Urine sample
pro-IAPP | 12 weeks
  Blood sample
IAPP (Islet Amiloide Polipeptide) | 12 weeks
  Boold sample

SECONDARY OUTCOMES:
Short-chain fatty acids profiling | 12 weeks
  Blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Regina Menezes, PhD, Principal Investigator — Lusofona University - CBIOS
Locations (1):
- Lusofona University, Lisbon, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stumvoll M, Goldstein BJ, van Haeften TW. Type 2 diabetes: principles of pathogenesis and therapy. Lancet. 2005 Apr 9-15;365(9467):1333-46. doi: 10.1016/S0140-6736(05)61032-X. PMID 15823385
- [Background] Raimundo AF, Ferreira S, Tomas-Barberan FA, Santos CN, Menezes R. Urolithins: Diet-Derived Bioavailable Metabolites to Tackle Diabetes. Nutrients. 2021 Nov 27;13(12):4285. doi: 10.3390/nu13124285. PMID 34959837
- [Background] Banihani SA, Makahleh SM, El-Akawi Z, Al-Fashtaki RA, Khabour OF, Gharibeh MY, Saadah NA, Al-Hashimi FH, Al-Khasieb NJ. Fresh pomegranate juice ameliorates insulin resistance, enhances beta-cell function, and decreases fasting serum glucose in type 2 diabetic patients. Nutr Res. 2014 Oct;34(10):862-7. doi: 10.1016/j.nutres.2014.08.003. Epub 2014 Aug 20. PMID 25223711
- [Background] Mansoor K, Bardees R, Alkhawaja B, Mallah E, AbuQatouseh L, Schmidt M, Matalka K. Impact of Pomegranate Juice on the Pharmacokinetics of CYP3A4- and CYP2C9-Mediated Drugs Metabolism: A Preclinical and Clinical Review. Molecules. 2023 Feb 24;28(5):2117. doi: 10.3390/molecules28052117. PMID 36903363
- [Background] Raimundo AF, Ferreira S, Pobre V, Lopes-da-Silva M, Brito JA, Dos Santos DJVA, Saraiva N, Dos Santos CN, Menezes R. Urolithin B: Two-way attack on IAPP proteotoxicity with implications for diabetes. Front Endocrinol (Lausanne). 2022 Dec 15;13:1008418. doi: 10.3389/fendo.2022.1008418. eCollection 2022. PMID 36589826